CLINICAL TRIAL: NCT03776149
Title: Therapeutic Role of Dietary Nitrates on Cardiovascular Function in Cancer Survivors Treated With Anthracycline Chemotherapy
Brief Title: Cardiovascular Function in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Carl Ade, M.S., Ph.D., Assistant Professor, Kansas State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro9264
Record Dates: First submitted 2018-05-14; First posted 2018-12-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cancer Survivor With History of Anthracycline Chemotherapy

STUDY DESIGN:
Intervention Model Description: This study utilizes a 7-day randomized, double-blind, placebo-controlled crossover study design, in which individuals are initially supplemented with a nitrate-rich supplement in the form of a specifically formulated beetroot juice, or nitrate-poor placebo. Individuals will then entered a 7-day washout period before entering the opposing arm of the study.
Who Masked: Participant, Investigator
Masking Description: The supplement and placebo will be distributed to the individual by a member of the research team who is not involved with data collection or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (dietary nitrate) (Experimental): Over the 7 days preceding each testing session, participants will consume 140 ml per day of beetroot juice (Beet It (HeartBeet Ltd.), Ipswich, UK). During this time participants will be asked to abstain from use of antiseptic mouthwash as this has been shown to temporarily kill the bacteria that facilitate the reduction of nitrate to nitrite. All participants will be asked to refrain from consuming any antioxidant (e.g., Vit E or Fish Oil) supplements during the course of the study as these may impact the study findings.
  Interventions: Dietary Supplement: Beetroot juice
- Black currant juice (placebo control) (Placebo Comparator): Over the 7 days preceding each testing session, participants will consume 140 ml per day of a nitrate-depleted placebo. During this time participants will be asked to abstain from use of antiseptic mouthwash as this has been shown to temporarily kill the bacteria that facilitate the reduction of nitrate to nitrite. All participants will be asked to refrain from consuming any antioxidant (e.g., Vit E or Fish Oil) supplements during the course of the study as these may impact the study findings.
  Interventions: Dietary Supplement: Black currant juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Following randomization on day 1, subjects will consume either the nitrate or nitrate-free beverage for 7 days with outcome measurements performed on day 7. Following a 7 day washout, subjects will then consume the crossover beverage for 7 days with outcome measures performed on day 21.
  Arms: Beetroot juice (dietary nitrate)
Dietary Supplement: Black currant juice — Following randomization on day 1, subjects will consume either the nitrate or nitrate-free beverage for 7 days with outcome measurements performed on day 7. Following a 7 day washout, subjects will then consume the crossover beverage for 7 days with outcome measures performed on day 21.
  Arms: Black currant juice (placebo control)

SUMMARY:
The aim of the current project is to understand the effect of dietary nitrates (via beet-root juice), on its ability to improve parameters of cardiovascular health in cancer survivors with a history of anthracycline chemotherapy.

DETAILED DESCRIPTION:
Cancer remains one of the leading causes of death in modern society, but due in part to increasing rates of detection coupled with advanced therapies, of the ≈230,000 people newly diagnosed with breast cancer each year, approximately 90% are expected to live beyond 5 years. Despite the trend in improved cancer-related mortality, breast cancer survivors are at a significantly increased risk for cardiovascular disease (CVD) morbidity and mortality. As such the American Heart Association has recently highlighted the immediate need to evaluate changes in cardiovascular health and function in the early stages of cancer treatment.

The mechanisms of adjuvant therapies on cardiovascular function may be the result of increased generation of reactive oxygen species (ROS) and altered redox status, specifically the balance between nitric oxide and superoxide. As such, nitrate supplementation has been shown to attenuate Doxorubicin (chemotherapy drug)-induced ventricular function in animal models. These data implicate dietary nitrates as one potential therapeutic intervention that could be used to improve cardiovascular health in cancer survivors.

Beetroot juice (BRJ) is a nutritional supplement that has been studied to examine potential effects of dietary nitrates affecting vasodilation. The increased nitrate levels have been implicated in helping increase nitric oxide bioavailability, which have been shown to improve cardiovascular function in older adults and those with known cardiovascular disease. The question, however, of whether or not BRJ will enhance cardiovascular function in breast cancer survivors is yet to be determined.

The primary aim of the current investigation is to test the hypothesis that dietary nitrate supplementation, via beet-root juice, improves parameters of cardiovascular health in cancer survivors with a history of anthracycline chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* cancer survivors (at least 1 year post treatment)
* Prior administration of anthracycline chemotherapy
* partial/complete remission

Exclusion Criteria:

* Unable to provide informed consent
* Kidney disease
* High risk of kidney stones
* Diagnosed hemochromatosis
* Pregnant, breast feeding, or planning to become pregnant
* Non-English speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Left ventricular function | The change between day 1 and day 21
  Left ventricular function as measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Change in Vascular function | The change between day 1 and day 21
  Vascular function measured as changes in arterial stiffness and endothelial function.
Change in Blood pressure | The change between day 1 and day 21
  Local limb blood pressure measured in millimeters of mercury (mmHg) following study interventions/arms

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas State University - Clinical Integrative Physiology Laboratory, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patnaik JL, Byers T, DiGuiseppi C, Dabelea D, Denberg TD. Cardiovascular disease competes with breast cancer as the leading cause of death for older females diagnosed with breast cancer: a retrospective cohort study. Breast Cancer Res. 2011 Jun 20;13(3):R64. doi: 10.1186/bcr2901. PMID 21689398
- [Background] Mulrooney DA, Blaes AH, Duprez D. Vascular injury in cancer survivors. J Cardiovasc Transl Res. 2012 Jun;5(3):287-95. doi: 10.1007/s12265-012-9358-7. Epub 2012 Mar 29. PMID 22456863
- [Background] Chaosuwannakit N, D'Agostino R Jr, Hamilton CA, Lane KS, Ntim WO, Lawrence J, Melin SA, Ellis LR, Torti FM, Little WC, Hundley WG. Aortic stiffness increases upon receipt of anthracycline chemotherapy. J Clin Oncol. 2010 Jan 1;28(1):166-72. doi: 10.1200/JCO.2009.23.8527. Epub 2009 Nov 9. PMID 19901105
- [Background] Duquaine D, Hirsch GA, Chakrabarti A, Han Z, Kehrer C, Brook R, Joseph J, Schott A, Kalyanaraman B, Vasquez-Vivar J, Rajagopalan S. Rapid-onset endothelial dysfunction with adriamycin: evidence for a dysfunctional nitric oxide synthase. Vasc Med. 2003 May;8(2):101-7. doi: 10.1191/1358863x03vm476oa. PMID 14518612